CLINICAL TRIAL: NCT07366021
Title: The Effect of Comfort Care Packages Applied to Intensive Care Patients on Patients' Comfort Level and Physiological Parameters
Brief Title: Comfort Care Bundle
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: Tarsus University (Other); Halic University (Other); Uludag University (Other); Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Banu Terzi, Dr., Akdeniz University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TBAEK-354
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: ICU; Comfort; Bundle Care; Nursing Care; Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-Behavioral (Experimental): Comfort Care Bundle Contents:
  * Ensure and maintain Physical Comfort (Prevent and manage pain, support daily living activities)
  * Ensure and maintain Psychospiritual Comfort (Manage agitation-sedation and delirium)
  * Ensure and maintain Environmental Comfort (Arrange the environment to facilitate the patient's adaptation)
  * Ensure and maintain Sociocultural Comfort (Enable and maintain the patient's interaction with their environment, ensure family participation in care)
  Interventions: Behavioral: Comfort Care Bundle
- Routine ICU care group (No Intervention): To avoid negatively impacting the data collection environment in the research (preventing issues such as bias by the nurse performing the procedure, ethical dilemmas, etc.), the study will begin with the collection of data from a control group. The control group will receive routine nursing care from the clinic.

INTERVENTIONS:
Behavioral: Comfort Care Bundle — A multicomponent comfort care bundle consisting of physical, psychosocial, environmental, and sociocultural comfort interventions delivered by ICU nurses to enhance patient comfort and reduce discomfort.
  Arms: Intervention-Behavioral

SUMMARY:
Intensive care units (ICUs) are specialized units where numerous complex treatment and care procedures are applied. In these units, critically ill patients are exposed to stressful conditions and experience significant pain and other discomforts stemming from multiple internal and external factors that can alter their quality of life and trigger symptoms of post-traumatic stress disorder (PTSD). These discomforts can have various short-term or long-term consequences for patients after discharge from the ICU, such as anxiety and/or depression or PTSD, which can affect their quality of life. Therefore, knowing the negative factors affecting patient comfort in the ICU, as well as measuring patient comfort and eliminating or reducing these factors through comfort care, is crucial in reducing morbidity and mortality rates in patients. It is noteworthy that there is no specific care package in the literature aimed at improving ICU-specific comfort. Accordingly, this study aims to develop a "Comfort Care Package" to improve the comfort level of ICU patients. The research population will consist of all patients aged 18-65 years admitted to the intensive care units of Bursa City Hospital. This study will test the effect of the developed "Comfort Care Package" on the comfort level and physiological parameters of 88 ICU patients (control group=44 and study group=44) who meet the inclusion criteria and whose data were calculated using the G*Power 3.1 program. The study will begin with the collection of data from the control group. This group will receive routine ICU care. The study group will receive the Comfort Care Package. It is anticipated that the ICU-specific comfort care package developed within the scope of this study will make significant contributions to the creation of nursing care plans aimed at increasing the comfort levels of critically ill individuals. Therefore, in patients with improved comfort, targeted recovery outcomes may increase, mortality rates may decrease, and thus public health may be sustained.

ELIGIBILITY:
Inclusion Criteria:

* Staying in the intensive care unit for at least 48 hours
* Communication language being Turkish
* For non-intubated patients, GCS > 12; for intubated patients, GCS > 10 + intubated (verbal response)

Exclusion Criteria:

* Hearing and hearing problems
* History or diagnosis of cognitive impairment, mental illness, nervous system disorders, brain injury
* RASS score >1
* Delirium
* Admitted with a diagnosis of alcohol/drug intoxication
* Pregnant
* Hemodynamically unstable patients receiving high-dose inotropic/vasopressor drug therapy
* Transfer to another ICU
* Emergency discharge from the ICU for any reason

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
The Comfort Behaviors Checklist | O. Day and 7. Day
  The Comfort Behaviors Checklist consists of 30 behavioral indicators. In addition, Kolcaba suggests that if listening comfort is the sole measurement tool, the individual should digitally score their pain and comfort, and that comfort should also be evaluated using a lens. Listening is coded in 42 different ways: 2, 3, 5, 7, 8, 9, 11, 12, 13, 19, 20, 21, 22, 24, 25, 27. The list is scored on a 4-point Likert scale. Parts of the list that are unsuitable for people are listed with a score of 0. The total number of questions answered is multiplied by 4 to obtain the possible score. The terminology questions are translated, and the scores of all questions are taken into account to obtain the raw comfort score. Finally, the possible comfort scores are divided by the raw scores to obtain a decimal number. The decimal part of the resulting score is expressed as a two-digit number. Higher scores indicate a high level of comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] • Lynn, M. R. 1986. "Determination and quantification of content validity", Nursing Research, 35(6), 381-5. • Ma, P., Liu, J., Xi, X., Du, B., Yuan, X., Lin, H., Wang, Y., Su, J., Zeng, L. 2010. "Practice of sedation and the perception of discomfort during mechanical ventilation in Chinese intensive care units", Journal of Critical Care, 25, 451-457. • Malinowski, A., Stamler, L. L. 2002. "Nursing theory and concept development or analysıs. Comfort: exploration of the concept in nursing", Journal of Advanced Nursing, 39(6), 599-606. • Matthews, E. E. 2011. "Sleep disturbances and fatigue in critically ill patients", American Association of Critical Care Nurses Advanced Critical Care, 22(3), 204-224. • Misak, C. J. 2004. "The critical care experience", American Journal of Respiratory and Critical Care Medicine, 170, 357-359. • Olausson, S., Fridh, I., Lindahl, B., Torkildsby, A. B. 2019. "The Meaning of comfort in the intensive care unit", Crit Care Nurs Q, 42(3), 329-341. • Orçan, F. 2018. "Açımlayıcı ve doğrulayıcı faktör analizi: ilk hangisi kullanılmalı?", Eğitimde ve Psikolojide Ölçme ve Değerlendirme Dergisi, 9(4), 413-421. • Özkan, F., Şahinoğlu, A. H. 2009. "Ondokuz Mayıs Üniversitesi Tıp Fakültesi cerrahi yoğun bakım ünitesinde yatan 967 hastanın retrospektif analizi", Journal of Experimental Clinical Medicine, 26, 62-67. • Park, M. S., Kang, K. J., Jang, S. J., Lee, J. Y., Chang, S. J. 2018. "Evaluating test-retest reliability in patient-reported outcome measures for older people: A systematic review", Int J Nurs Stud., 79, 58-69. doi:10.1016/j.ijnurstu.2017.11.003. • Polat, M.G. 2007. "Yoğun bakımda fizyoterapi uygulamaları", Yoğun Bakım Dergisi, 7(3), 357-361. • Pugh, R. J. 2007. "The impact of noise in the intensive care unit", Critical and Emergency Care, 4, 12-18. • Riker, R. R., Picard, J. T., Fraser, G. L. 1999. "Prospective evaluation of the Sedation-Agitation Scale for adult critically ill patients", Crit Care Med, 27(7), 1325-132. • Şahin, M. G.,